CLINICAL TRIAL: NCT03089736
Title: Pain Related to Head and Neck Cancer (HNC); Implementation and Evaluation of Self-care Measure Due to the Same Illness During Radiotherapy (RT)
Brief Title: Pain Related to Head and Neck Cancer (HNC); Implementation and Evaluation of Self-care Measure Due to the Same Illness
Acronym: HNC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Bjorn Gerdle, Professor MD, Linkoeping University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HNC, pain-coaching during RT
Record Dates: First submitted 2015-08-26; First posted 2017-03-24 (Actual); Last update posted 2017-03-30 (Actual); Status verified 2017-03

CONDITIONS: Pain; Head and Neck Cancer
Keywords: Pain; Head and neck cancer; depression; anxiety; health; catastrophizing
MeSH Terms: conditions — Pain; Head and Neck Neoplasms; Depression; Anxiety Disorders | interventions — Educational Status; Self Care; Therapeutics

STUDY DESIGN:
Masking Description: All patients who referred to the Pain and Rehabilitation Centre at the University Hospital, asked about participation in the study. Of those who agreed to participate every second patient were distributed to the control group versus intervention group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TAU + Education and self care (Experimental): Treatment as usual (TAU; i.e. pharmacological treatments and advices) + structured education + instructions on self care
  Interventions: Behavioral: Education; Behavioral: Self Care; Other: Treatment as usual (TAU)
- Treatment as usual (TAU) (Other): Treatment as usual (TAU; i.e. pharmacological treatments and advices)
  Interventions: Other: Treatment as usual (TAU)

INTERVENTIONS:
Behavioral: Education — Six education areas was offered: pain and pain physiology, pain medication, side effects and prevention of side effects, abuse of medications, sleep advice and advice on anxiety.
  Arms: TAU + Education and self care
Behavioral: Self Care — The following instructions on self-care for pain relief: apply ice or crushed ice in the oral cavity, lubricating and antiseptic mouth rinses, pain relieving gel, tongue movements and gaps exercises. Prevention of dryness in the mouth and throat; saliva stimulants and saliva substitute agents in different preparations, increased measures of good oral hygiene. Physical activities and regular rest once to several times per day. Sleep restriction and measures to treat sleep disorders.
  Arms: TAU + Education and self care
Other: Treatment as usual (TAU) — pharmacological treatment + advices

SUMMARY:
The purpose of this study is to evaluate the effect of individual education and individual self-care measures on pain intensity, perceived health, mood and sleep during and after treatment with radiotherapy for head and neck cancer.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the effect of individual education and individual self-care measures on pain intensity, perceived health, mood and sleep during and after treatment with radiotherapy for head and neck cancer

ELIGIBILITY:
Inclusion Criteria:

All HNC patients who went through RT and were referred to the Pain and Rehabilitation Centre at the University Hospital (Linköping, Sweden) were invited to participate in the study which run from January 2015 - March 2017.

-

Exclusion Criteria:

Non Swedish speaking individuals, severe social and/or psychological disorders, severe cognitive conditions,other serious medical conditions.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2017-03-19 (Actual)

PRIMARY OUTCOMES:
Change in Pain intensity | Change from baseline pain intensity at 20 weeks
  Pain intensity the actual day using a numeric rating scale.
Change in Pain Interference | Change from baseline pain interference at 20 weeks
  Pain interference the actual day using a numeric rating scale
Change in Perceived health index | Change from baseline EQ-5D index at 20 weeks
  Perceived health according to the index based on five dimensions of European Quality of Life instrument (EQ-5D index)
Change in Perceived health scale | Change from baseline EQ-VAS at 20 weeks
  Perceived health according to the visual analgue scale of European Quality of Life instrument (EQ-VAS)

SECONDARY OUTCOMES:
Change in depression | Change from baseline depression at 20 weeks
  Depression scale of Hospital and Depression Scale (HADS)
Change in anxiety | Change from baseline anxiety at 20 weeks
  Anxiety scale of Hospital and Depression Scale (HADS)
Change in catastrophizing | Change from baseline catastrophizing at 20 weeks
  Total score of Pain Catastrophizing scale

CONTACTS AND LOCATIONS:
Overall Officials: Bjorn Gerdle, Professor MD, Principal Investigator — Rehabilitation Medicine, Linkoeping University

IPD SHARING:
Plan to Share IPD: No